CLINICAL TRIAL: NCT03316677
Title: Intraoperative Testing of Colorectal Anastomosis - Air or Water (Methylene Blue)?
Acronym: ITCORA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMC11261-16CTIL
Record Dates: First submitted 2017-01-15; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-01

CONDITIONS: ColoRectal Cancer; Colonic Diverticulitis; Anastomotic Leak; Anastomotic Complication; Anastomosis
Keywords: anastomotic leak; colorectal; anastomosis testing; Intraoperative testing
MeSH Terms: conditions — Colorectal Neoplasms; Diverticulitis, Colonic; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- colorectal resection and anastamosis (Other): Intraoperative testing of colorectal anastomoses
  1. Insert a Foley catheter through the anus into the rectum.
  2. Insufflate the Foley balloon with 5 cc of air.
  3. fill the pelvic space with 500 CC of warm saline
  4. Insufflate air into the rectum up to a pressure of 35 mmH2o as measured by external manometer
  5. Remove the saline from the pelvic space.
  6. Inject methylene blue in to the rectum up to a pressure of 35 mmH2o measured by external manometer
  7. Remove the methylene blue from rectum.
  NB the above procedures are standard practice for assessing the quality of colorectal anastomoses during colorectal surgery.
  The purpose of the study is to compare these standard methods of evaluation to determinant which method is superior
  Interventions: Procedure: Intraoperative testing of colorectal anastomoses; Procedure: Stapled colorectal anastomoses

INTERVENTIONS:
Procedure: Intraoperative testing of colorectal anastomoses — 1. Insert a Foley catheter through the anus into the rectum.
  2. Insufflate the Foley balloon with 5 cc of air.
  3. Air tight leak test with saline and insufflating air: fill the pelvic space with 500 CC of warm saline
  4. Insufflate air into the rectum up to a pressure of 35 mmH2o as measured by external manometer
  5. Remove the saline from the pelvic space.
  6. Inject diluted dye (methylene blue) in to the rectum up to a pressure of 35 mmH2o measured by external manometer
  7. Remove the methylene blue from rectum.
  NB the above procedures are standard practice for assessing the quality of colorectal anastomoses during colorectal surgery.
  The purpose of the study is to compare these standard methods of evaluation to determinant which method is superior
Procedure: Stapled colorectal anastomoses — After the resection we do the stapled colorectal anastomosis with a standard circular stapler as part of the regular procedure

SUMMARY:
A leak from a colorectal anastomosis is a post-operative complication surgeons fear the most, following colonic resection. Over the years, there have been multiple suggestions for intraoperative tests for the integrity of the colorectal anastomosis.

Two of the most common tests that are performed routinely are:

1. Air tight leak test - filling the pelvis with saline and insufflating air trans anal - looking for air bubbles in the saline filled pelvis.
2. Injecting diluted dye (methylene blue) trans anal, and looking for blue dye stains on gauze pads covering the outer side of anastomosis.

The aim of the study is to compare the two methods, and to assess if there is a superior method. A secondary aim is to establish standards to perform the test, mainly to assess the appropriate pressure to apply on the anastomosis.

In this prospective study patients scheduled to undergo colonic resection of their distal part of the colon/ rectum with colorectal anastomosis, will have both testing methods performed sequentially and will be followed post-operative to assess the yield and sensitivity of the testing methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 undergoing elective colonic resection of their distal part of the colon/ rectum with colorectal anastomosis in a laparoscopic or open approach for a benign or malignant colonic disease.

Exclusion Criteria:

* Emergent colonic resections,
* Colonic resections with no colorectal anastamosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
the predictive value of intraoperative anastomosis testing on anastomotic leak. | 30 days
  The presence or absence of a post-operative clinical anastomotic leak

SECONDARY OUTCOMES:
The sensitivity of the 2 methods of intraoperative anastomosis testing. | Both findings will be obvious (if present) immediately after the test is performed
  We will compare the occurence of air leak with the occurence of methylene blue leak in each patient

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Avital, MD, Principal Investigator — Meir Medical Center, Israel

REFERENCES:
- [Derived] Rudnicki Y, White I, Tiomkin V, Lahav L, Raguan B, Avital S. Intraoperative evaluation of colorectal anastomotic integrity: a comparison of air leak and dye leak tests. Tech Coloproctol. 2021 Jul;25(7):841-847. doi: 10.1007/s10151-021-02453-4. Epub 2021 Apr 27. PMID 33905010